CLINICAL TRIAL: NCT00387452
Title: Exercise and Cardiovascular Control During Upright Tilt in Older Adults With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Kenneth Madden, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H04-70001; ORSIL# 05-0820
Record Dates: First submitted 2006-10-11; First posted 2006-10-13 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Cardiovascular; Diabetic
Keywords: Aging; Type 2 diabetes; exercise; aerobic training; strength training; glucose metabolism arterial baroreceptors; heart rate variability; cerebral autoregulation; tilt table study; transcranial Doppler; autonomic nervous system
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (Active Comparator)
  Interventions: Behavioral: Aerobic Exercise and Strength Exercise
- 2 (Active Comparator)
  Interventions: Behavioral: Strength training
- 3 (No Intervention): No intervention, only testing during 6 months.

INTERVENTIONS:
Behavioral: Aerobic Exercise and Strength Exercise — 6 months of aerobic training exercise. regulated by heart rate; work up to 80% of maximal heart rate on treadmill or stationary bike; 3 hours a week, 90% attendance.
  Arms: 1
Behavioral: Strength training — 6 months of strength training exercise using weight machines involving legs and arms: 12-15 repetitions of weights per exercise; 3 hours a week, 90% attendance.
  Arms: 2

SUMMARY:
Older persons with diabetes have a harder time maintaining blood pressure when standing up. When blood pressure drops when standing up, fainting may occur. This study will see how regular exercise can improve the ability of the body to keep blood pressure up when standing. We want to see how this improvement varies with different types of exercise. The types of exercise that we will be studying are aerobic (running or cycling on a stationary bike) and strength training (weight lifting).

DETAILED DESCRIPTION:
1. PURPOSE: Older adults with diabetes faint frequently, due to an impairment in the cardiovascular control mechanisms (arterial baroreceptor function, autonomic nervous system function and cerebral autoregulation) that prevent syncope. The purpose of this study is to examine the ability of different intensities of aerobic exercise to reverse these impairments.
2. HYPOTHESES: a) Aerobic or strength training will improve the compensatory cardiovascular responses that prevent syncope in older adults with Type 2 diabetes. Aerobic training will:

   * increase arterial baroreflex sensitivity
   * increase heart rate variability (marker of autonomic nervous system function)
   * decrease cerebrovascular resistance
   * improve cerebral autoregulation during upright tilt. b) There will be relationship between the improvement in compensatory cardiovascular responses and aerobic or strength training.

     c) The majority of the benefits of aerobic or strength exercise on the above parameters will with which training, allowing for the design of more practicable training prescriptions than that used in a research setting.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 5 years treated with diet alone or oral agents Nonsmoker for at least 5 years Subjects must be sedentary BMI between 24 and 35 All subjects will have a fasting glucose of <12 mM and a hemoglobin A1c < 8.5% All subjects must have developed hypertension CDA guidelines (systolic greater than 130 or diastolic greater than 80)

Exclusion Criteria:

* Abnormalities on complete blood count, electrolytes or creatinine, on resting ECG, treadmill exercise stress test Significant pulmonary, exercise-limiting orthopedic or neurological impairment Evidence of valvular disease, exercise-induced syncope, angina, arrhythmias or peripheral vascular disease Poor blood pressure control as defined as systolic blood pressure greater than or equal to 160 mm Hg or diastolic blood pressure greater than or equal to 90 mm Hg Total cholesterol/HDL cholesterol greater than or equal to 5.0 or LDL cholesterol greater than or equal to 4.21 mmol/L Peripheral neuropathy severe enough to cause discomfort (for safety reasons) Significant orthostatic hypotension defined as a drop in systolic blood pressure greater than 30 mmHg during one of five consecutive arterial blood pressure readings immediately after changing position from lying to standing for safety.

Overt diabetic nephropathy excluding subjects with a urine albumin to creatinine ratio of greater than 2.0 in men or 2.8 in women Diabetic retinopathy

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 64 (Actual)
Dates: Start 2006-02 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Pulse wave velocity (central and peripheral)
Drop in middle cerebral artery velocity with upright tilting
Drop in blood pressure with upright tilt
Arterial baroreflex sensitivity
Time and frequency domain measures of heart rate variability

SECONDARY OUTCOMES:
Fasting blood glucose, HgbA1C
VO2max
Dynamometry measures of muscle strength
Resting and maximal heart rate
Waist to hip ratio, BMI
Lean body mass/% fat
Catecholamines
Increase in Gosling's pulsatility index
Linear transfer-function analysis of cerebral autoregulation during upright tilt

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Madden, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital Research Pavilion, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No